CLINICAL TRIAL: NCT06568744
Title: Fluid Intolerance Signals as Safety Limits to Prevent Fluid-induced Harm During Septic Shock Resuscitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220607015; 1230475 (Other Grant/Funding Number: ANID FONDECYT)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: Septic Shock
Keywords: fluid overload; resuscitation; capillary refill time; POCUS
MeSH Terms: conditions — Shock, Septic; Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will follow a resuscitation algorithm aimed at macrohemodynamic stabilization and improvement of tissue hypoperfusion. Fluid administration will be tailored according to fluid responsiveness status, fluid intolerance signals, and hypoperfusion signals such as capillary refill time. Mechanical ventilation and sedation will follow standard management as per current recommendations.
  Interventions: Other: Intervention resuscitation
- Standard of Care (Active Comparator): This group will follow a resuscitation algorithm aimed at macrohemodynamic stabilization and improvement of tissue hypoperfusion. Fluid administration will be tailored according to fluid responsiveness status, and hypoperfusion signals such as capillary refill time. Mechanical ventilation and sedation will follow standard management as per current recommendations.
  Interventions: Other: Standard of Care resuscitation

INTERVENTIONS:
Other: Intervention resuscitation — In fluid responsive patients, fluid intolerance will be checked.
  Lung Ultrasound (LUS): Anterior LUS with 4-point assessment at each hemithorax. Min:0 and a max:24. Low risk: < 10; intermediate risk: 10-14 or delta of 2 points. High risk: >14, or an increase >4 from baseline.
  VExUS: Low risk: Grade 0-1. Intermediate risk: 2. High risk: 3 E/e' ratio: Low risk: <8. Intermediate risk: 8-13. High risk >14. Central venous pressure (CVP): Low risk <12 mmHg. Intermediate risk: 12-15 mmHg or a delta of 3 mmHg. High risk > 15 mmHg or >5 mmHg increase after a fluid challenge.
  In low-risk, a fluid challenge of 500 ml of balanced crystalloid will be performed in 30 minutes. If intermediate risk, a fluid challenge of 250 ml of balanced crystalloid in 30 minutes. If high-risk signals, alternative strategies (vasopressor and inodilator tests) will be deployed. After each challenge, peripheral perfusion, fluid responsiveness and intolerance will be re-assessed.
  Arms: Intervention
Other: Standard of Care resuscitation — In fluid responsive patients, fluid challenges of 500 ml of balanced crystalloid will be performed in 30 minutes. After a fluid challenge, peripheral perfusion status and fluid responsiveness will be re-measured. If the patient persists with hypoperfusion, successive fluid challenges will be performed until hypoperfusion resolves or the patient becomes fluid unresponsive. If hypoperfusion signals persists and the patient becomes fluid unresponsive, alternative resuscitation interventions will be deployed, which include: 1) vasopressor titration to higher mean arterial pressure (MAP) targets in a MAP-test, and 2) addition of an inotrope to increase cardiac output in an inodilator test. If hypoperfusion fails to resolve, rescue therapies such as high-volume hemofiltration will be initiated.
  Arms: Standard of Care

SUMMARY:
The goal of this multicentric randomized controlled trial is to compare, in septic shock patients who require further fluid resuscitation, two strategies of administering fluids. The intervention group will integrate fluid intolerance signals to the decision making process, while the control group will follow standard of care, for a 6 hour study protocol. The main question it aims to answer is

1. To compare the effect of both resuscitation strategies on fluid-induced harm, assessed by the change in pulmonary, cardiac, and renal function biomarkers during the study period.
2. To assess the safety of both resuscitation strategies on hypoperfusion resolution, measured by the improvement of capillary refill time (CRT) and lactate during the study period.
3. To determine the dynamics of the different fluid intolerance signals

DETAILED DESCRIPTION:
Fluids are the first-line hemodynamic therapy during septic shock resuscitation, restoring tissue perfusion by effectively increasing cardiac output and oxygen delivery. Nevertheless, resuscitation fluids can be seen as a double-edged sword since they have a narrow therapeutic index. In the one hand, insufficient fluid administration can perpetuate hypoperfusion, leading to irreversible tissue hypoxia, while excessive fluid administration can lead to fluid-induced harm. The extreme scenario of this condition, fluid overload, has been consistently associated with worse clinical outcomes, including increased risks of prolonged mechanical ventilation, acute kidney injury and mortality. As an eminently retrospective diagnosis, it may underestimate the importance of timely recognition of fluid-induced harm during the resuscitation period and could shift clinicians' efforts to treatment rather than prevention. Thus, identifying organ-specific venous congestion signals early on during the resuscitation process is desirable and could avoid these adverse outcomes. Recent studies have shown that venous congestion signals are present even during the first day of ICU admission.

The investigators hypothesized that in critically ill patients with septic shock, a fluid resuscitation strategy that integrates fluid intolerance signals as safety limits will prevent fluid-induced harm, without compromising hypoperfusion resolution, compared to a standard resuscitation strategy.

To confirm this hypothesis, the investigators propose a multicenter prospective randomized controlled study in 62 critically ill patients with septic shock, comparing two strategies for conducting fluid resuscitation, aiming to decrease fluid-induced harm. One strategy will follow the standard of care, while the other will rest on real-time ultrasound-based monitoring of fluid intolerance signals. The latter approach will allow clinicians to limit fluid administration when potentially deleterious signals appear. The impact of both strategies on fluid-induced harm will be assessed by the evolution of key organ function biomarkers, namely lungs, heart, and kidneys during the 6-hour study period. Perfusion dynamics will be assessed by capillary refill time and arterial lactate kinetics during the study period. Patients will receive general monitoring and management according to ICU standards. Patients will be followed-up for 28 days for other relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed or suspected septic shock
* < 24 hours since diagnosis
* Hypoperfusion signal (altered arterial lactate or CRT) that requires further resuscitation
* Mechanical ventilation
* Positive fluid responsiveness status

Exclusion Criteria:

* Pregnancy
* Do-not-resuscitate status
* Acute coronary syndrome
* Active bleeding
* Severe concomitant acute respiratory distress syndrome (ARDS) (PaO2:FiO2 ratio < 100)
* Anticipated surgery, prone positioning, or renal replacement therapy in the next 6 hours
* Refractory shock according to attending physician
* BMI > 40.
* Inadequate echocardiographic window

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Delta of PaO2: fraction of inspired oxygen (FiO2) ratio between 0-6 hours | 6 hours
  evolution of lung function during the study period (6h)

SECONDARY OUTCOMES:
Delta of proBNP between 0-6 hours | 6 hours
  evolution of cardiac function during the study period (6h)
Delta of plasma neutrophil gelatinase-associated lipocalin (NGAL) between 0-6 hours | 6 hours
  evolution of renal function during the study period (6h)
Delta of creatinine between 0-6 hours | 6 hours
  evolution of renal function during the study period (6h)
Delta of capillary refill time between 0-6 hours | 6 hours
  evolution of peripheral perfusion during the study period (6h)
Delta of arterial lactate between 0-6 hours | 6 hours
  evolution of lactate during the study period (6h)

OTHER OUTCOMES:
Delta of PaO2:FiO2 ratio between 24 hours | 24 hours
  lung function at the first day since recruitment
Delta of plasma NGAL between 0-24 hours | 24 hours
  evolution of kidney function during the first day since recruitment
Delta of creatinine between 0-24 hours | 24 hours
  evolution of kidney function during the first day since recruitment
Delta of proBNP between 0-24 hours | 24 hours
  evolution of cardiac function during the first day since recruitment
Delta of arterial lactate between 0-24 hours | 24 hours
  evolution of lactate during the first day since recruitment
Delta of capillary refill time between 0-24h | 24 hours
  evolution of peripheral perfusion during the first day since recruitment
Fluid balance at 24 hours | 24 hours
  fluids administered during the first day of protocol
Mortality | 28 days
  mortality rate during the first 28 days
ICU length of stay | 28 days
  length of stay in the intensive care unit
Organ dysfunction free days | 28 days
  days alive without vasopressor, renal replacement or mechanical ventilation support

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Kattan, MD, PhD, Principal Investigator — Pontifiia Universidad Catolica de Chile
Locations (3):
- Chile (3):
  - Hospital Biprovincial Quillota-Petorca, Quillota
  - Hospital Barros Luco, Santiago
  - Hospital Clinico UC Christus, Santiago

IPD SHARING:
Plan to Share IPD: Yes
data sharing will be anonymized upon reasonable request to the corresponding author
Supporting Information: Study Protocol, CSR
Time Frame: After study completion
Access Criteria: upon reasonable request to the PI.

REFERENCES:
- [Background] Munoz F, Born P, Bruna M, Ulloa R, Gonzalez C, Philp V, Mondaca R, Blanco JP, Valenzuela ED, Retamal J, Miralles F, Wendel-Garcia PD, Ospina-Tascon GA, Castro R, Rola P, Bakker J, Hernandez G, Kattan E. Coexistence of a fluid responsive state and venous congestion signals in critically ill patients: a multicenter observational proof-of-concept study. Crit Care. 2024 Feb 19;28(1):52. doi: 10.1186/s13054-024-04834-1. PMID 38374167
- [Background] Kenny JS, Prager R, Rola P, Haycock K, Basmaji J, Hernandez G. Unifying Fluid Responsiveness and Tolerance With Physiology: A Dynamic Interpretation of the Diamond-Forrester Classification. Crit Care Explor. 2023 Dec 12;5(12):e1022. doi: 10.1097/CCE.0000000000001022. eCollection 2023 Dec. PMID 38094087
- [Background] Kattan E, Castro R, Miralles-Aguiar F, Hernandez G, Rola P. The emerging concept of fluid tolerance: A position paper. J Crit Care. 2022 Oct;71:154070. doi: 10.1016/j.jcrc.2022.154070. Epub 2022 Jun 2. PMID 35660844
- [Background] Kattan E, Ospina-Tascon GA, Teboul JL, Castro R, Cecconi M, Ferri G, Bakker J, Hernandez G; ANDROMEDA-SHOCK Investigators. Systematic assessment of fluid responsiveness during early septic shock resuscitation: secondary analysis of the ANDROMEDA-SHOCK trial. Crit Care. 2020 Jan 23;24(1):23. doi: 10.1186/s13054-020-2732-y. PMID 31973735
- [Background] Zampieri FG, Damiani LP, Bakker J, Ospina-Tascon GA, Castro R, Cavalcanti AB, Hernandez G. Effects of a Resuscitation Strategy Targeting Peripheral Perfusion Status versus Serum Lactate Levels among Patients with Septic Shock. A Bayesian Reanalysis of the ANDROMEDA-SHOCK Trial. Am J Respir Crit Care Med. 2020 Feb 15;201(4):423-429. doi: 10.1164/rccm.201905-0968OC. PMID 31574228
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Bagshaw SM, Brophy PD, Cruz D, Ronco C. Fluid balance as a biomarker: impact of fluid overload on outcome in critically ill patients with acute kidney injury. Crit Care. 2008;12(4):169. doi: 10.1186/cc6948. Epub 2008 Jul 24. PMID 18671831